# **Informed Consent Form**

## Research title:

Effects of Expressive Writing on Stress and Work-Related Outcomes among Student Nurse Interns: a randomized controlled trial

# NCT ID:

Not yet assigned

## Date of the document:

October 17th, 2023

### Informed Consent Form

Dear prospective participants:

My team would like to invite you to participate in a study exploring the effects of a writing intervention on clinical practice experience and feelings. The following is an explanation of the research project, including information on the purpose, significance, and specific research protocol, and you can ask the project leader any project-related questions (Project leader: **Ji Xuan**; phone no.: +86 17835856131; email: **jixuan0101@163.com**). Please read this informed consent form carefully and make your decision to participate in the study carefully.

This study aims to investigate the effects of an intervention program based on a writing format on undergraduate student nurse interns' clinical practice experience and feelings. Participants will be instructed to write (15 minutes twice a week for ten weeks) and fill in the questionnaires (one day before the intervention, one day after the intervention, and four weeks, eight weeks, and 12 weeks after the end of the intervention).

Writing about unpleasant experiences may induce negative emotions; if they are more severe, you can always stop writing for emotional calming and contact our team psychologist if necessary.

If you want to find out exactly how this program works, you need to follow these rules:

- Cooperate with the writing task based on the instructions;
- Complete the related questionnaires.

We guarantee:

- All your data will be kept confidential but only be identified with a code for this study;
- Participation is entirely voluntary, and you may withdraw from this study at any time,
  even if you have signed the informed consent form.

If you have read this Informed Consent Form, understand the study, and would like to participate in this study, please sign below.

| Signi |
|-------|
| Date. |